CLINICAL TRIAL: NCT05762081
Title: The Effect of Two Different Bed Baths Applied to Patients on Mechanical Ventilation Support on Vital Signs: A Randomized Controlled Trial
Brief Title: The Effect of Two Different Bed Baths Applied to Patients on Mechanical Ventilation Support
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Sercan Kara, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-282
Record Dates: First submitted 2023-02-02; First posted 2023-03-09 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-02

CONDITIONS: The Effect of Two Different Bed Baths; Patients on Mechanical Ventilation Support
Keywords: Nursing; Mechanical Ventilation; Baths; Vital Sings

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Individuals who have undergone wiping bathing with disposable wipes
  Interventions: Procedure: Disposable Wipes for wiping baths
- Control Group (Sham Comparator): Individualswho have undergone bathing with a traditional bath
  Interventions: Procedure: Traditional bed bath

INTERVENTIONS:
Procedure: Disposable Wipes for wiping baths — A disposable wipe bath is a type of bath that is applied to bed-bound or unconscious patients and weak individuals by wiping the entire body.
  Arms: Intervention Group
Procedure: Traditional bed bath — Traditional bed bathing is a type of bathing applied to bed-bound or unconscious patients and weak individuals by wiping the entire body with soap and water.
  Arms: Control Group

SUMMARY:
The aim of this study was to determine the effect of two different methods (traditional bed bathing and disposable antibacterial wipe bathing) on vital signs in patients on mechanical ventilation support.

DETAILED DESCRIPTION:
The study is planned as a randomized controlled study to determine the effect of the performance of two types of bed (bed-traditional and disposable antibacterial wipe bath) on respiratory parameters and vital signs in adult patients with different clinical conditions connected to mechanical ventilation. At the end of the study, it is aimed to evaluate the effect of traditional and disposable antibacterial wiping baths on vital signs in patients on mechanical ventilation support.

Relatives of the patients who meet the inclusion criteria will be informed about the purpose, content and method of the study and the sample group (experimental and control) will be formed by obtaining written permission from those who voluntarily agree to participate in the study. Determination of the experimental and control groups will be provided by https://www.randomizer.org/ website. The wiping bath protocol with disposable antibacterial wipes will be applied to the experimental group in accordance with the literature, and the traditional bed bath protocol will be applied to the patients in the control group by the researcher himself. Patient Information Form containing information about the demographic characteristics and medical status of the patients included in the study; vital signs (pulse, systolic and diastolic blood pressure, body temperature, respiratory rate and SpO2) and blood gas data will be recorded 3 times in total (before the bath - current blood gas value, immediately after the bath - morning routine blood gas, 30 minutes or more after the bath - the first blood gas taken with the physician's order) based on the values in the routine blood gas measurements of the clinic, partial arterial oxygen and partial arterial carbon dioxide parameters will be recorded in the vital signs follow-up form. All data collection tools will be completed by the researcher himself.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older, whose voluntary consent is obtained from a relative or legal guardian,
* Dependent on mechanical ventilation,
* Not receiving antihypertensive and sedation therapy,
* Not taking inotropic drugs that directly affect vital signs (esmolol, noradrenaline dopamine, adrenaline, dopamine nitrate, etc.),
* No wound that prevents bathing,
* Moving it does not cause any problems,
* Minimum 24 hours in intensive care,
* Patients with blood gas readings taken 30 minutes or more after bathing

Exclusion Criteria:

* Not dependent on mechanical ventilation,
* Receiving antihypertensive and sedation therapy,
* Taking inotropic drugs that directly affect vital signs (esmolol, noradrenaline dopamine, adrenaline, dopamine nitrate, etc.),
* A person with a wound that prevents bathing,
* It is important to note that moving it does not cause any problems,
* Less than 24 hours in intensive care,
* Patients in whom blood gas readings were not taken 30 minutes or more after bathing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-08-15 (Estimated); Study Completion 2023-11-15 (Estimated)

PRIMARY OUTCOMES:
Change in Blood Pressure | Baseline and immediately after bathing, 30 minutes after bathing
  Blood pressure will be measured on the patient monitor. Results will be reported in mmHg.
Change in Pulse Rate | Baseline and immediately after bathing, 30 minutes after bathing
  Pulse rate will be measured on the patient monitor. The results presented as beat per minute.
Change in Respiratory Rate | Baseline and immediately after bathing, 30 minutes after bathing
  Respiratory rate will be measured on the patient monitor. Higher scores mean a worse result.
Change in Body Temperature | Baseline and immediately after bathing, 30 minutes after bathing
  A calibrated non-contact infrared thermometer will be used to measure body temperature. Results will be reported in Celcius.
Change in Oxygen Saturation | Baseline and immediately after bathing, 30 minutes after bathing
  Oxygen Saturation will be measured on the patient monitor. Approaching %100 is concidered positive. Higher scores mean a better result.
Change in Score of Acute Physiology and Chronic Health Evaluation II (APACHE II). | Baseline and immediately after bathing, 30 minutes after bathing
  Score of Acute Physiology and Chronic Health Evaluation II (APACHE II).
Change in Mechanical Ventilation Mode | Baseline and immediately after bathing, 30 minutes after bathing
  The patient's mechanical ventilation mode will be observed. SIMV, CBAP, etc.
Change in Partial Oxygen Pressure (PaO2) | Baseline and immediately after bathing, 30 minutes after bathing
  The level of partial oxygen pressure is measured as mmHg in arterial blood gase analysis
Change in Partial Carbon Dioxide Pressure | Baseline and immediately after bathing, 30 minutes after bathing
  Change in the partial carbon dioxide pressure in the arterial blood (blood gas analysis) at a defined oxygen flow rate (L/min)

CONTACTS AND LOCATIONS:
Locations (1):
- Sercan KARA, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Aydın, A. (2011). Kişisel Hijyen ve Yatak Yapımı. İçinde T. Aştı ve A. Karadağ (Ed.). Klinik Uygulama Becerileri ve Yöntemleri. Adana: Nobel Tıp Kitabevi; (375-462).
- [Background] Coyer FM, O'Sullivan J, Cadman N. The provision of patient personal hygiene in the intensive care unit: a descriptive exploratory study of bed-bathing practice. Aust Crit Care. 2011 Aug;24(3):198-209. doi: 10.1016/j.aucc.2010.08.001. Epub 2010 Sep 15. PMID 20829060
- [Background] EI-Soussi AH, Asfour Hl.( 2016). Examining bed-bath practices ofcritically ill patients. J Nurs Educ Practice .;( 12):1-11. doi : https: / /doi.org/10 .5430/ jnep.v6n12pl.
- [Background] Garrido D, Assioun JJ, Keshishyan A, Sanchez-Gonzalez MA, Goubran B. Respiratory Rate Variability as a Prognostic Factor in Hospitalized Patients Transferred to the Intensive Care Unit. Cureus. 2018 Jan 23;10(1):e2100. doi: 10.7759/cureus.2100. PMID 29581913
- [Background] Groven FM, Zwakhalen SM, Odekerken-Schroder G, Joosten EJ, Hamers JP. How does washing without water perform compared to the traditional bed bath: a systematic review. BMC Geriatr. 2017 Jan 25;17(1):31. doi: 10.1186/s12877-017-0425-4. PMID 28118815
- [Background] Kızıl, H.(2015). Mekanik Ventilasyonda Olan Entübe Çocuklara Uygulanan Yatak Banyosunun Yaşam Bulgularına Ve Oksijen Satürasyonuna Etkileri. Yüksek Lisans Tezi. Marmara Üniversitesi Sağlık Bilimleri Enstitüsü. İstanbul
- [Background] Moller G, Magalhaes AMM (2015). Bed baths: nursing staff workload and patient safety. Texto Contexto Enferm.;24(4) :1044-52. doi : http ://d x .doi. org/10.1590/ 0104-0707201500003110014.
- [Background] Oz O, Uysal G, Duzkaya DS. Effect of Two Bathing Methods on Physiologic Parameters in Pediatric Intensive Care. Clin Nurs Res. 2022 Jun;31(5):858-865. doi: 10.1177/10547738211043337. Epub 2021 Sep 18. PMID 34538125
- [Background] Paulela DC, Bocchi SC, Mondelli AL, Martin LC, Regina A.(2018) Sobrinho. Effecti veness of bag bath on microbial load: clinical trial. Acta Paul Enferm . ;31(1) :7-16. doi: http://dx.doi.org/10.1590/1982-0194201800003
- [Background] Quiroz S, Castro C, Tirado AF, Rodriguez LM . (2012)Alteraciones hemodinamicas del paciente critico card iovascular durante larealizaci6n del bafio diario. Medicina UPB. https://redib.org/Record/oai_articulo1202311- modelo-de-adaptaci%C3%B3n-de-roy-en-el-ba%C3%B1o-en-cama erişim:04.06.2022
- [Background] Silva LF, Miranda AFA, Silva FVF, Rabelo ACS, Almeida PC, Ponte KMA. (2014) Vital signs and nursing procedures in postoperative period of cardiac surgery. J Nurs UFPE on line.; 8(3):719-25 . doi: 10.5205/reuol.5149-42141-1- SM .0803201429
- [Background] Skewes SM. Skin care rituals that do more harm than good. Am J Nurs. 1996 Oct;96(10):33-5. No abstract available. PMID 8863646
- [Background] Şendir, M., ve Büyükyılmaz, F. (2014). Yoğun Bakım Ünitesinde Çalışan Hemşirelerin İki Farklı Yatak Banyosu Uygulamasına Ilişkin Görüşleri: YarıKalitatif Çalışma ve Maliyet Analizi. 19-22 Kasım 2014 3. Temel Hemşirelik Bakımı Kongresi Bildiri Kitabı, 19-22 Kasım, Antalya.
- [Background] Şendir,M..(2012). Hemşirelik Esasları Uygulama Rehberi. İçinde T. Aştı ve A. Karadağ (Eds.), Kişsel Temizlik ve Giyinme Aktivitesi (2. cilt). İstanbul: İstanbul Kitapevleri ve Yayıncılık;275-279.
- [Background] Tai CH, Hsieh TC, Lee RP. The Effect of Two Bed Bath Practices in Cost and Vital Signs of Critically Ill Patients. Int J Environ Res Public Health. 2021 Jan 19;18(2):816. doi: 10.3390/ijerph18020816. PMID 33477909
- [Background] Taylor, C.R., Lillis, C., LeMone, P. and Lynn, P. (2011). Fundamentals of nursing (7thed). US: Lippincott Williams &Wilkins
- [Background] Toledo LV, Salgado PO, Souza CC, Brinati LM, Januario CF, Ercole FF. Effects of dry and traditional bed bathing on respiratory parameters: a randomized pilot study. Rev Lat Am Enfermagem. 2020;28:e3264. doi: 10.1590/1518-8345.3668.3264. Epub 2020 Jun 1. PMID 32491124
- [Background] Uludağ, S.(2022). Yoğun Bakım Hastalarında İki Banyo Yönteminin Yaşam Bulguları Ve Oksijen Satürasyonu Üzerine Etkisi. Yüksek Lisans Tezi. Marmara Üniversitesi Sağlık Bilimleri Enstitüsü. İstanbul
- [Background] Ünsal, A.(2013). Hijyen Uygulamaları. İçinde T. Aştı ve A. Karadağ (Eds.), Hemşirelik Esasları Hemşirelik Bilimi ve Sanatı (2. cilt). İstanbul: Akademi Basım ve Yayıncılık;446-465.
- [Background] Zaybak, A. ve Güneş, Ü. (2009). Yatağa bağımlı hastalarda yatak banyosunun yaşam bulgularına etkisi. Atatürk Üniversitesi Hemşirelik Yüksekokulu Dergisi, 12(4), 91-95.